

| TEMPLATE: EXEMPT RESEARCH INFORMATION SHEET | |
|---------------------------------------------|--------------|
| NUMBER | VERSION DATE |
| HRP-UT926 | 9/13/2024 |

#### **Research Information Sheet**

#### **Basic Study Information**

**Title of the Project:** Adapting Stress First Aid (SFA) to the needs of Harm Reduction Workers (HRWs) serving Persons Who Use Drugs (PWUD) – Training and Pilot Testing Phase (Aim 2 and Aim 3)

**UT Austin Investigator:** Suzannah Creech, PhD, Dell Medical School, The University of Texas at Austin

## Invitation to Voluntarily Participate in a Research Study

You are invited to be part of a research study. Your participation is voluntary and it is totally up to you to decide whether you want to participate. Even if you decide to be part of the study now, you may change your mind and stop at any time.

# What is the study about and why are we doing it?

This research project is focusing on supporting the well-being of the harm reduction workforce including Harm Reduction, Community Health and Peer support Workers who do harm reduction work with persons who use drugs. We collaborated with both harm reduction workers and leaders at harm reduction organizations to adapt an existing support program aimed at reducing occupational stress. With your help, we have the unique opportunity to pilot and test the feasibility, acceptability, and effectiveness of adapted Stress First Aid (SFA) for Harm Reduction Workers materials utilizing team support champions, to inform change for the harm reduction workforce across the country.

## What will happen if you take part in this study?

If you agree to take part in this study, you will be asked to participate in a 4-month field test of the feasibility, acceptability and appropriateness of SFA for Harm Reduction Workers (HRWs). You will participate in a virtual 2-hour team support champion facilitated SFA training and up to 4, 30-minute virtual monthly learning collaborative meetings that will introduce SFA concepts and how to use SFA on a day-to-day basis in your work life and with coworkers. The team support champions are workers in harm reduction, like you, that will lead you in the 2-hour training to introduce you to SFA and its principles and lead you, as the participants, in the monthly learning collaborative meetings. Other members of our team, trained in SFA, will lead trainings and collaboratives as needed. The trainings and monthly learning collaborative meetings will not be recorded. You will complete a baseline assessment prior to the SFA training, two follow-ups at 2 and 4 months after baseline, and a brief post-training questionnaire and an optional reaction interview (approximately 1-hour total for assessments and 30 minutes for an audio and/or video-recorded Zoom interview). The same survey will be used at baseline and for the two follow-up assessments. Your email will be linked to your survey responses only for purposes of facilitating follow-up and pairing your baseline, 2-month, and 4-month follow-up assessments. After the follow-up assessment period has passed, the research team will remove your email from your survey responses. You will be asked questions about social support,



burnout, use of the SFA practices, job-related well-being, secondary traumatic stress, coping strategies, confidence in managing certain situations, work engagement, and turnover. If interviewed, you will be asked about your reactions to the Stress First Aid curriculum. We expect that this study will take about **5-5.5 hours of your time**.

# **Contact Information for the Study Team**

If you have any questions, concerns, or complaints about this research now or in the future, you may contact the following:

Anmol Desai, MPH and Juliette Rau, MSW Program Coordinators Email: SFA@austin.utexas.edu

# Contact Information for Questions about Your Rights as a Research Participant

If you have questions about your rights as a research participant, or wish to obtain information, ask questions, or discuss any concerns about this study with someone other than the researcher(s), please contact the following:

The University of Texas at Austin Institutional Review Board

Phone: 512-232-1543

Email: irb@austin.utexas.edu

#### Compensation

To thank you for your time and participation, you will receive \$50 gift card for completing each full assessment and \$25 for the post-intervention assessment/interview, for a total of \$175. If you withdraw before the end of the study, you will receive a \$50 gift card for each full assessment completed. You will be responsible for any taxes assessed on the compensation.

Payment received as compensation for participation in research is considered taxable income to the research subject. If payment to an individual is equal to or exceeds \$600 in any one calendar year, The University of Texas at Austin is required to report this information to the Internal Revenue Service (IRS). If the compensation you receive from participation in this research in combination with all other compensation received from The University of Texas at Austin is equal to or exceeds \$600 in the current calendar year, you must provide IRS 1099 related information.

#### **Required Disclosures**

Under certain situations, we may break confidentiality. If during the study we learn about [child abuse or neglect, or that someone is a clear, serious, and direct harm to self or others,] we will report this information to the appropriate authorities [including the police and/or the Texas Department of Family and Protective Services, and/or emergency medical facility.]

To help protect your privacy, this research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They



also cannot provide information, documents, or samples that may identify you as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state, or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop sponsoring United Sates federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers, or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.